CLINICAL TRIAL: NCT03970304
Title: CVD 37000: Immunity and Microbiome Studies at Intestinal and Systemic Sites in Ty21a Vaccinated Adults
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Bruce Greenwald, Professor of Medicine, University of Maryland, Baltimore
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HP-00056321
Record Dates: First submitted 2019-05-29; First posted 2019-05-31 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Typhoid Vaccination

STUDY DESIGN:
Intervention Model Description: Volunteers who choose to take part in this study will receive the licensed FDA approved Oral Typhoid Vaccine (Vivotif). Volunteers also have the possibility of being a control participant who will not be vaccinated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Vaccination, Colonoscopy (Experimental): Individuals receive immunization with Vivotif typhoid vaccine prior to routine colonoscopy examination. During colonoscopy, small bowel biopsies will be obtained to examine immune responses and microbiota at the mucosal level; brushings will also be obtained.
  Interventions: Drug: Vivotif Typhoid Oral Vaccine
- Colonoscopy, Vacciniation, Colonoscopy (Experimental): Individuals receive immunization with Vivotif typhoid vaccine after initial colonoscopy exam and specimen collection and prior to a routine follow up colonoscopy examination during which additional specimens will be collected.
  Interventions: Drug: Vivotif Typhoid Oral Vaccine
- Colonoscopy Without Vaccination (No Intervention): Individuals do not receive immunization but consent to collection of specimens during colonoscopy. The specimens to be collected in all three groups include stool, saliva, and small bowel biopsies (terminal ileum).

INTERVENTIONS:
Drug: Vivotif Typhoid Oral Vaccine — The 4 doses (1 capsule each) will be administered on alternate days, e.g., days 0, 2, 4, and 7 (± 1 day) under the supervision of the study coordinator(s).
  Other Names: Ty21a Typhoid Oral Vaccine
  Arms: Colonoscopy, Vacciniation, Colonoscopy; Vaccination, Colonoscopy

SUMMARY:
This is an open-label, non-randomized study. The purpose of this study is to better understand how vaccines against typhoid fever affect the normal immune system and bacteria in the intestine. Patients having standard-of-care colonoscopies will be divided into 3 groups:

Group 1: Vivotif typhoid vaccination then colonoscopy; Group 2: Colonoscopy, then Vivotif typhoid vaccination, then follow-up colonoscopy; Group 3: Colonoscopy without vaccination.

The Vivotif typhoid vaccine used in this study is licensed by the Food and Drug Administration (FDA) for travelers to developing countries. Volunteers will be asked to donate tissue, blood, saliva and stool samples for studying how the body responds to the typhoid vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Undergoing colonoscopy for screening or surveillance for colorectal cancer at the University of Maryland
* Provide written informed consent prior to initiation of any study procedures
* Healthy, as defined by considered fit to undergo outpatient elective colonoscopy by the referring health care provider

Exclusion Criteria:

* Pregnancy or nursing mother
* Known coagulopathy or bleeding disorder preventing mucosal biopsy
* History of Crohn's disease or ulcerative colitis
* Surgical removal of the ileocecal valve or any part of the small or large intestine
* Allergic reaction to oral typhoid vaccine in the past
* Immunosuppression from illness or treatment, including

  * immune-deficiency disorders such as Human Immunodeficiency Virus (HIV) or Acquired Immunodeficiency Syndrome (AIDS)
  * leukemia, lymphoma, or cancers
  * immune suppressive medications or treatments, such as corticosteroids or radiation
* Receipt of any other vaccine two weeks prior to receipt of Ty21a
* Positive urine pregnancy test (HCG) prior to colonoscopy or vaccination

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2013-10-24 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of Responders | approximately 5 years
  Percentage of responders by cytokine production (Interferon-gamma (IFN-gamma) or Tumor Necrosis Factor-alpha (TNF-α)) by mass cytometry or flow cytometry. Responders will be defined as those volunteers showing increases post-immunization of >0.1% of positive CD8+ cells for IFN-gamma or TNF-α over baseline (pre-immunization) values.) or Tumor Necrosis Factor-alpha (TNF-α)) by mass cytometry or flow cytometry.

CONTACTS AND LOCATIONS:
Locations (1):
- Universtiy of Maryland, Baltimore, Center for Vaccine Development and Global Health, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Booth JS, Goldberg E, Patil SA, Barnes RS, Greenwald BD, Sztein MB. Age-dependency of terminal ileum tissue resident memory T cell responsiveness profiles to S. Typhi following oral Ty21a immunization in humans. Immun Ageing. 2021 Apr 19;18(1):19. doi: 10.1186/s12979-021-00227-y. PMID 33874975
- [Derived] Booth JS, Goldberg E, Barnes RS, Greenwald BD, Sztein MB. Oral typhoid vaccine Ty21a elicits antigen-specific resident memory CD4+ T cells in the human terminal ileum lamina propria and epithelial compartments. J Transl Med. 2020 Feb 25;18(1):102. doi: 10.1186/s12967-020-02263-6. PMID 32098623